CLINICAL TRIAL: NCT00847210
Title: A Phase 1, Randomized, Open-Label, Parallel Group, Multicenter Study to Evaluate the Pharmacokinetics and Safety of Dexlansoprazole Modified Release Capsules (30 mg and 60 mg) in Adolescents With Symptomatic Gastroesophageal Reflux Disease
Brief Title: Pharmacokinetic and Safety of Dexlansoprazole in Adolescents With Gastroesophageal Reflux Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T-P107-163; U1111-1114-1891 (Registry Identifier: WHO)
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Results first posted 2010-10-05 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Gastroesophageal Reflux
Keywords: Esophageal Reflux; Gastro-Esophageal Reflux; Gastroesophageal Reflux Disease; GERD; Regurgitation, Gastric; Heartburn; Drug Therapy; Adolescent
MeSH Terms: conditions — Gastroesophageal Reflux; Laryngopharyngeal Reflux; Heartburn | interventions — Dexlansoprazole; Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexlansoprazole MR 30 mg QD (Experimental)
  Interventions: Drug: Dexlansoprazole MR
- Dexlansoprazole MR 60 mg QD (Experimental)
  Interventions: Drug: Dexlansoprazole MR

INTERVENTIONS:
Drug: Dexlansoprazole MR — Dexlansoprazole MR 30 mg, capsules, orally, once daily for up to 7 days.
  Other Names: TAK-390MR; Kapidex; Dexilant
  Arms: Dexlansoprazole MR 30 mg QD
Drug: Dexlansoprazole MR — Dexlansoprazole MR 60 mg, capsules, orally, once daily for up to 7 days.
  Other Names: TAK-390MR; Kapidex; Dexilant
  Arms: Dexlansoprazole MR 60 mg QD

SUMMARY:
The purpose of this study is to asses the pharmacokinetics and safety of dexlansoprazole modified release (MR), once daily (QD), in adolescent subjects (age 12-17 years old) with Symptomatic Gastroesophageal Reflux Disease.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease is a condition of multifactorial etiology resulting in the reflux of gastric contents into the esophagus through the lower esophageal sphincter. The prevalence of Gastroesophageal reflux disease in the pediatric population is becoming increasingly recognized and documented. It is a chronic disease that can persist through adulthood with symptoms in older children and adolescents being similar to those seen in adults. The prevalence of gastroesophageal reflux disease increases with age, from 2.5% of children between the ages of 3 and 9 years, to 8.5% of those between the ages of 10 and 17 years.

Younger children generally present with extra-esophageal manifestations, regurgitation, and epigastric pain, while older children and adolescents typically present with adult-type gastroesophageal reflux disease symptoms of heartburn and regurgitation. Treatment for gastroesophageal reflux disease is aimed at alleviating symptoms and healing the esophageal inflammation.

This study evaluated the pharmacokinetics and safety of dexlansoprazole MR in the pediatric population (ages 12-17) and determined if the pharmacokinetic profile is similar to that in adults given the same dose.

ELIGIBILITY:
Inclusion Criteria:

* Body weight is greater than or equal to 30 kg.
* Females of childbearing potential who are sexually active must agree to use an acceptable form of contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Must have an estimated creatinine clearance greater than or equal to 80 mL/minute as determined from the Cockcroft-Gault formula.
* Participants who take prescription or non-prescription proton pump inhibitors, histamine receptor antagonists (except cimetidine), sucralfate, or antacids on a regular or as required basis must agree to discontinue usage throughout the study.
* Must have a history of gastroesophageal reflux disease symptoms, as documented by a physician, for at least 2 months prior to Screening or is currently symptomatic.
* Must be able to swallow study drug capsule or must be able to ingest study drug granules sprinkled on 1 tablespoon of applesauce.

Exclusion Criteria:

* Has evidence of current cardiovascular, central nervous system, hepatic, hematopoietic, renal, or metabolic dysfunction, serious allergy, asthma, or allergic skin rash.
* Has any finding in his/her medical history, physical examination, or safety clinical laboratory tests giving reasonable suspicion of a disease that might interfere with the conduct of the trial or that would contraindicate taking dexlansoprazole MR or a similar drug in the same class.
* Has a known hypersensitivity to any proton pump inhibitors or any component of the formulation of dexlansoprazole MR (see most current version of the Investigator Brochures).
* Has a history of malignant disease.
* Has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody.
* Has a known history of infection with the human immunodeficiency virus.
* Has donated or lost greater than or equal to 300 mL blood volume, undergone plasmapheresis, or has had a transfusion of any blood product within 90 days prior to the first dose of study drug.
* Is required to take or intends to continue taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication.
* Has consumed grapefruit or grapefruit juice within 14 days prior to the first dose of study drug or is unwilling to agree to abstain from grapefruit or grapefruit juice while participating in the study.
* Has a history of alcohol abuse or illegal drug use or drug abuse in the past, or tests positive for alcohol or drugs of abuse at the initial Screening Visit or Day -1 or is unwilling to agree to abstain from alcohol and drugs throughout the study.
* Has used a product containing nicotine within 90 days prior to the first dose of study drug or has a positive cotinine screen at the initial Screening Visit or Day -1 or is unwilling to agree to abstain throughout the study.
* Has participated in a study of an investigational agent (including dosing or follow up) within 30 days prior to first dose of study drug.
* Has an initial Screening Visit or Day -1 laboratory value that the principal investigator considers to be clinically significant.
* Participant is determined to be a CYP2C19 isozyme poor metabolizer (ie, genotyped homozygous non-wild type).
* Is unlikely to comply with the protocol or is unsuitable for any other reason per the opinion of the investigator

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Pharmacovigilance, Study Director — Takeda
Locations (3):
- United States (3):
  - Anaheim, California
  - Cypress, California
  - Overland Park, Kansas

REFERENCES:
- [Result] Kukulka M, Wu J, Perez MC. Pharmacokinetics and safety of dexlansoprazole MR in adolescents with symptomatic GERD. J Pediatr Gastroenterol Nutr. 2012 Jan;54(1):41-7. doi: 10.1097/MPG.0b013e31822a323a. PMID 21716130
- See also: Dexilant Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=9efb34b3-fb69-4190-a2be-a90b8cb94e25&filetypecode=DEXILANTPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 3 investigative sites in the United States from 31 May 2009 to 10 September 2009.
Pre-assignment Details: Participants were enrolled in one of two, dexlansoprazole modified release (MR), once-daily (QD) treatment groups. 100% of participants randomized completed this study.
Groups:
- Dexlansoprazole MR 30 mg QD: Dexlansoprazole MR 30 mg, capsules, orally, once daily for up to 7 days.
- Dexlansoprazole MR 60 mg QD: Dexlansoprazole MR 60 mg, capsules, orally, once daily for up to 7 days.
Period: Overall Study
Arm/Group | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD | Total
Number analyzed (Participants) | 18 | 18 | 36
Age Continuous [Mean (Standard Deviation); unit: years] | 14.6 (1.65) | 14.6 (1.89) | 14.6 (1.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) Pharmacokinetic Parameter
Description: Tmax: Time to reach the Maximum Plasma Concentration (Cmax), equal to time (hours) to Cmax, as observed on Day 7.
Time Frame: After 7 days of dosing.
Population: All participants who had Tmax estimated were included in the analysis for this parameter. One participant in the 30 mg group was excluded from the pharmacokinetic (PK) analysis because most of the PK samples were not collected, and hence no PK parameters were estimable. There was no imputation for missing values.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Number analyzed (Participants) | 17 | 18
hours | 4.65 (2.909) | 3.31 (1.519)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 30 mg QD vs Dexlansoprazole MR 60 mg QD; This study was not powered for any hypothesis testing. For Tmax, an analysis of variance (ANOVA) model was fitted that included fixed effect of age group, regimen and interaction of age group and regimen. If the interaction term was not statistically significant, it was not included in the final model. The site effect was also tested in the model, and was not included in the final model if it was not statistically significant (P>0.05). Pairwise comparisons between regimens were conducted; Test type: Superiority or Other; p = 0.095, ANOVA — There was no statistical significant difference (p-value >0.05) in Tmax between the 30 mg and 60 mg dose group. Both age group and site did not have statistically significant effects on Tmax

2. Primary Outcome: Cmax: Maximum Observed Plasma Concentration Pharmacokinetic Parameter.
Description: Maximum Observed Plasma Concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: After 7 days of dosing.
Population: All participants who had Cmax estimated were included in the analysis for this parameter. One participant in the 30 mg group was excluded from the PK analysis because most of the PK samples were not collected, and hence no PK parameters were estimable. There was no imputation for missing values.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Number analyzed (Participants) | 17 | 18
ng/mL | 691 (367.5) | 1136 (582.2)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 30 mg QD vs Dexlansoprazole MR 60 mg QD; This study was not powered for any hypothesis testing. For natural logarithm of dose-normalized Cmax, an ANOVA model was fitted that included fixed effect of age group, regimen and interaction of age group and regimen. If the interaction term was not statistically significant, it was not included in the final model. Site effect was tested in the model, and was not included in the final model if not statistically significant (P>0.05). Pairwise comparisons between regimens were conducted; Test type: Superiority or Other; p = 0.289, ANOVA; ratio of the central values for Cmax = 1.210, 90% CI 2-sided [0.897 to 1.630] — Ninety percent confidence intervals for assessing the dose proportionality of dexlansoprazole pharmacokinetics between regimens were computed based on the frame work of ANOVA

3. Primary Outcome: AUC(0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration Pharmacokinetic Parameter.
Description: Area Under the Plasma Concentration Versus Time Curve (AUC(0-tlqc)) is a measure of total plasma exposure to the drug from Time 0 to Time of the Last Quantifiable Concentration (AUC[0-tlqc]).
Time Frame: After 7 days of dosing.
Population: All participants who had AUC(0-tlqc) estimated were included in the analysis for this parameter. One participant in the 30 mg group was excluded from the PK analysis because most of the PK samples were not collected, and hence no PK parameters were estimable. There was no imputation for missing values.
Measure: Mean (Standard Deviation); unit: ng*hr/mL/mg
Arm/Group | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Number analyzed (Participants) | 17 | 18
ng*hr/mL/mg | 2842.32 (1313.827) | 5113.72 (2987.508)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 30 mg QD vs Dexlansoprazole MR 60 mg QD; This study was not powered for any hypothesis testing. For Tmax, an ANOVA model was fitted that included fixed effect of age group (12-14 years and 15 17 years), regimen and interaction of age group and regimen. If the interaction term was not statistically significant, it was not included in the final model. The site effect was also tested in the model, and was not included in the final model if it was not statistically significant (P>0.05). Pairwise comparisons between regimens were conducted; Test type: Superiority or Other; p = 0.402, ANOVA; Ratio of the dose-normalized AUC(0-tlqc) = 1.158, 90% CI 2-sided [0.864 to 1.551] — Ninety percent confidence intervals for assessing the dose proportionality of dexlansoprazole AUC(0-tlqc) between regimens were computed based on the frame work of ANOVA

4. Primary Outcome: AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours Postdose Pharmacokinetic Parameter.
Description: AUC(0-24) is measure of Area Under the Curve over the dosing interval (tau) (AUC(0-tau]), where tau is the length of the dosing interval - 24 hours in this study).
Time Frame: After 7 days of dosing.
Population: All participants who had AUC(0-24) estimated were included in the analysis for this parameter. One participant in the 30 mg group was excluded from the PK analysis because most of the PK samples were not collected, and hence no PK parameters were estimable. There was no imputation for missing values.
Measure: Mean (Standard Deviation); unit: ng*hr/mL/mg
Arm/Group | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Number analyzed (Participants) | 16 | 18
ng*hr/mL/mg | 2886.26 (1355.182) | 5119.81 (2986.453)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 30 mg QD vs Dexlansoprazole MR 60 mg QD; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.388, ANOVA; Ratio of the central values for dose-nor = 1.168, 90% CI 2-sided [0.864 to 1.579] — Ninety percent confidence intervals for assessing the dose proportionality of dexlansoprazole AUC(0-24) between regimens were computed based on the frame work of ANOVA

5. Primary Outcome: Terminal Phase Elimination Half-life (T1/2) Pharmacokinetic Parameter.
Description: Terminal Phase Elimination Half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Time Frame: After 7 days of dosing.
Population: All participants who had T1/2 estimated were included in the analysis for this parameter. One participant in the 30 mg group was excluded from the PK analysis because most of the PK samples were not collected, and hence no PK parameters were estimable. No statistical tests were performed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Number analyzed (Participants) | 16 | 18
hours | 1.66 (0.871) | 2.59 (1.379)

6. Primary Outcome: Oral Clearance (CL/F) Pharmacokinetic Parameter.
Description: CL/F is apparent clearance of the drug from the plasma, calculated as the drug dose divided AUC(0-24), expressed in L/hr.
Time Frame: After 7 days of dosing.
Population: All participants who had CL/F estimated were included in the analysis. One participant in the 30 mg group was excluded from the PK analysis because most of the PK samples were not collected, and hence no PK parameters were estimable. There was no imputation for missing values. No statistical tests were performed.
Measure: Mean (Standard Deviation); unit: liter/hr
Arm/Group | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Number analyzed (Participants) | 16 | 18
liter/hr | 12.81 (6.092) | 15.29 (7.524)

7. Primary Outcome: Terminal Elimination Rate Constant (λz) Pharmacokinetic Parameter.
Description: Terminal elimination rate constant (λz) is the rate at which drugs are eliminated from the body.
Time Frame: After 7 days of dosing.
Population: All participants who had λz estimated were included in the analysis. One participant in the 30 mg group was excluded from the PK analysis because most of the PK samples were not collected, and hence no PK parameters were estimable. There was no imputation for missing values. No statistical tests were performed.
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Number analyzed (Participants) | 16 | 18
1/hr | 0.5264 (0.25425) | 0.3404 (0.17406)

8. Primary Outcome: Apparent Volume of Distribution (Vz/F) Pharmacokinetic Parameter.
Description: Vz/F is the distribution of a drug between plasma and the rest of the body following oral administration, calculated as CL/F divided by λz.
Time Frame: After 7 days of dosing.
Population: All participants who had Vz/F estimated were included in the analysis for this parameter. One participant in the 30 mg group was excluded from the PK analysis because most of the PK samples were not collected, and hence no PK parameters were estimable. There was no imputation for missing values. No statistical tests were performed.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Number analyzed (Participants) | 16 | 18
L | 28.90 (21.208) | 58.50 (46.100)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are defined as those reported after the first dose and no more than 30 days after the last dose of study drug.
Description: There were no deaths, serious adverse events or significant adverse events during the study.
Arm/Group | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 7/18 | 5/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexlansoprazole MR 30 mg QD (N=18) | Dexlansoprazole MR 60 mg QD (N=18)
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Eructation (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2
Feelings of Body Temperature Change (General disorders) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Headache (Nervous system disorders) | 1 | 2
Dizziness (Nervous system disorders) | 1 | 1
Presyncope (Nervous system disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
For outcome measures #4, 5, 6, 7 and 8, outcomes could not be estimated for one participant in the 30 mg dose group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights therefrom or any data, information or materials obtained or generated in the performance of it's obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.